CLINICAL TRIAL: NCT03842410
Title: Solyx Single-Incision SlingDynamic Intraoperative Standing Sling Technique (DISST) as an Office-based Procedure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Michigan Institution of Women's Health PC (Other)
Responsible Party: Principal Investigator, Salil Khandwala, Director, Michigan Institution of Women's Health PC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ODISST
Record Dates: First submitted 2019-02-07; First posted 2019-02-15 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single-Incision Sling (Other): Intervention with in office solyx suburethral sling DISST
  Interventions: Device: Single-Incision Sling

INTERVENTIONS:
Device: Single-Incision Sling — Solyx Single-Incision Sling for correction of stress urinary incontinence done in the office.
  Other Names: Solyx Single-incision sling

SUMMARY:
This study will assess the feasibility and success of performing the SolyxTM SIMUS in the office using the Dynamic Interactive Standing Sling Technique (DISSTTM). Study endpoints will be feasibility, composite success, complications, and patient and physician acceptance.

DETAILED DESCRIPTION:
The single-incision midurethral sling (SIMUS) is a procedure where there are no exit incisions. There is a 15 mm suburethral incision with the sling being attached with anchors to the obturator muscle on each side. This procedure has potentially lesser side-effects compared to the longer slings however, the literature has not found the SIMUS to be as effective as the long slings. In our recently published study, the DISSTTM technique has significantly improved the success of the SIMUS procedure as the sling can be tested for proper application in vivo.

As we have performed several of these procedures in the operating room entirely under local anesthesia, we have decided to perform this procedure in an office setting using the same safety precautions as in a hospital operating room.

Performing this procedure in the office has significant benefits for the patient, the healthcare industry, and the economy overall. Moving away from a hospital setting has significant psychological benefits. This will increase patient acceptance and therefore will become appealing to many more women who may be shying away from treatment.

It would also eliminate the risk of nosocomial infections for the patient and family members, improve efficiency as the wait time would be negligible, and would reduce the expense of the entire treatment as hospital costs would not feature in the equation.

This study will assess the feasibility and success of performing the SolyxTM SIMUS in the office using the Dynamic Interactive Standing Sling Technique (DISSTTM). Study endpoints will be feasibility, composite success, complications, and patient and physician acceptance.

ELIGIBILITY:
Inclusion Criteria:

* SUI with hypermobility of the urethrovesical (UV) junction
* American Society of Anesthesiologists (ASA) classes I or II
* Ages ranging 21-89 years
* Have the ability to stand for CST during the procedure
* Have failed behavioral therapy
* Completed childbearing

Exclusion Criteria:

* ASA classes III or IV
* Need for concomitant surgery
* Poor compliance for office-based approach
* Demonstrate concomitant urgency incontinence on urodynamic testing

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-05-31 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Subject tolerability of the Solyx SIMUS in the office using the Dynamic Interactive Standing Sling Technique (DISST) | intraoperative
  Subject tolerability will be assessed using a 10-cm Visual Analogue Scale rating tolerability of the procedure. The Visual Analog Scale measures discomfort of the procedure with 0 being no discomfort and 10 being severe discomfort.
Surgeon difficulty of performing the Solyx SIMUS in the office using the Dynamic Interactive Standing Sling Technique (DISST) | intraoperative
  Surgeon difficulty will be determined by a 5-point Likert scale ranging from 1 (very easy) to 5 (very difficult).
Ability to achieve DISST SUCCESS | intraoperative
  Defined as a negative intraoperative standing cough stress test (CST) at bladder fullness.
Complications of performing the Solyx SIMUS in the office using the Dynamic Interactive Standing Sling Technique (DISST) | intraoperative
  Any intraoperative complications will be documented

SECONDARY OUTCOMES:
Improvement in overall urinary incontinence (stress and urge incontinence) | 3, 6, 12, 24 and 60 months post operative
  Subject will complete the Medical, Epidemiologic, and Social Aspects of Aging (MESA) urinary incontinence questionnaire to assess improvement in urge incontinence and stress incontinence. Subjects will also complete the Patient Global Impression of Improvement (PGI-I) questionnaire as it pertains to stress urinary incontinence.
Sexual function | 3, 6,12, 24 and 60 months post operative
  Subject will complete the Pelvic Organ Prolapse/Urinary Incontinence Sexual (PISQ-12) questionnaire to assess changes in sexual function.
Improvement in patient quality of life as it relates to urinary symptoms | 3, 6,12, 24 and 60 months post operative
  Subject will complete Incontinence Impact Questionnaire (IIQ-7) to assess changes in quality of life related to urinary symptoms.
Subject satisfaction with overall improvement from sling procedure | 3, 6, 12, 24 and 60 months post operative
  Subject will completed satisfaction questionnaire to determine patients overall satisfaction with the procedure and results
Post operative pain | pre-procedure to 7 days after procedure
  Post operative pain will be assessed using a McCarthy pain scale questionnaire, which ranges from "No Pain Sensation" to "Most Intense Pain Sensation Imaginable". Pain will be assessed at rest, during daily activities, during sex, lifting, or other strenuous work in the last 24 hours. This will be completed prior to surgery, the day of, and the 7 days following surgery.
Post operative complications | post procedure to 12, 24 and 60 months
  At post operative visits patients will be asked and assessed for post operative complications (based upon the Clavien Dindo classification)
Return to pre-surgical activities | Pre-procedure to return to 60 months
  Patients will be asked what activities they engage in prior to surgery including work, exercise, social, and household activities. At each post operative visit the patient will be asked when they returned to pre-surgical activities.

CONTACTS AND LOCATIONS:
Overall Officials: Salil Khandwala, M.D., Principal Investigator — Advanced Urogynecology of Michigan, P.C.
Locations (1):
- Advanced Urogynecology of Michigan P.C, Dearborn, Michigan, United States

IPD SHARING:
Plan to Share IPD: No